CLINICAL TRIAL: NCT03938766
Title: Upregulation of PSMA Receptors After Androgen Deprivation Therapy on PSMA PET/CT Imaging in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Gad Abikhzer, Principal Investigator, Jewish General Hospital
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CODIM-MDM-18-001
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PSMA PET/CT (Other): Repeat PSMA PET/CT after ADT
  Interventions: Diagnostic Test: PSMA PET/CT

INTERVENTIONS:
Diagnostic Test: PSMA PET/CT — Repeat PSMA PET/CT 4 weeks post initiation of clinically indicated ADT in patients with prior negative PSMA PET/CT performed for biochemical recurrence.

SUMMARY:
Prostate specific membrane antigen (PSMA) is a unique membrane bound glycoprotein, which is overexpressed on prostate cancer cells and is well-characterized as an imaging biomarker of prostate cancer. Studies have shown that PSMA PET/CT can detect prostate cancer lesions with excellent contrast and a high detection rate even when the level of prostate specific antigen is low. PSMA imaging is considered the gold standard in imaging of biochemical recurrence, with detection rate of recurrence in 79.5% of patients, in the largest series of 1007 patients. Despite these excellent results, there remains approximately 20% of patients in whom the site of biochemical recurrence cannot be identified and further research is needed into improving detection rates.

Androgen deprivation therapy (ADT), represents the standard of care treatment for most men with a rising serum PSA and no evidence of disseminated disease on imaging modalities. There has been some preliminary data that imaging patients early after initiation of ADT therapy may increase detection rates of recurrence sites.

The objective of this study is to evaluate if prostate cancer patients with biochemical recurrence and negative PSMA PET/CT can demonstrate in-vivo upregulation of PSMA receptors in an attempt to improve detection rates of recurrent prostate cancer. Patients who are started on ADT when clinically indicated, will have repeat PSMA PET/CT at 4 weeks following initiation of ADT therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 18 years or older
* Previous diagnosis of prostate cancer following radical prostatectomy or primary radiation therapy, with biochemical recurrence.
* Prior negative PSMA PET/CT within 2 months prior to study entry
* ECOG performance status 0 - 3, inclusive
* Able to understand and provide written informed consent
* Initiation of androgen deprivation therapy within 5 weeks prior to study PSMA PET/CT
* Able to tolerate the physical/logistical requirements of a PET/CT scan

Exclusion Criteria

* Medically unstable patients
* Patients who exceed the safe weight limit of the PET/CT bed (200 kg) or who cannot fit through the PET/CT bore (70 cm diameter)
* Patients with unmanageable claustrophobia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Detection rates of recurrence | 2 years
  The percentage of 18F-DCFPyL PET/CT positive for identification of biochemical recurrence sites in patients with prostate cancer following initiation of ADT therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No